CLINICAL TRIAL: NCT02818426
Title: Anticancer Therapeutic Vaccination Using Telomerase-derives Universal Cancer Peptides in Metastatic Non Small Cell Lung Cancer : A Phase I/II Study
Brief Title: Universal Cancer Peptide-based Vaccination in Metastatic NSCLC
Acronym: UCPVax
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Invectys (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCPVax; 2015-001712-35 (EudraCT Number)
Record Dates: First submitted 2016-05-20; First posted 2016-06-29 (Estimated); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Metastatic Non-small Cell Lung Cancer
Keywords: cancer immunotherapy; CD4 T lymphocyte helper; telomerase
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UCPVax (Experimental): UCPVax is a therapeutic cancer vaccine composed of two peptides called UCP2 and UCP4 derived from telomerase combined with Montanide ISA 51 VG as adjuvant.
  The two peptides UCP2 and UCP4 will be emulsified in Montanide ISA 51 and injected subcutaneously in separate sites (one site per peptide), at days 1, 8, 15, 29, 36 and 43 (priming phase) following by boost vaccination every 8 weeks for 12 months.
  Interventions: Drug: UCPVax

INTERVENTIONS:
Drug: UCPVax

SUMMARY:
UCPVAx is a therapeutic vaccine based on the telomerase-derived UCP designed to induce strong TH1 CD4 T cell responses in cancer patients.

Three doses of UCPVax (0,25 mg, 0,5 mg and 1 mg) will be tested in this phase I/II study by using Continuous Reassessment Method (CRML) dose escalation design model.

The phase I is a dose escalation study designed to evaluate safety of use of UCPVax and to estimate its Maximum Tolerated Dose (MTD).

The phase II is a dose deescalation designed to evaluate the immunogenicity of UCPVax according to the dose level.

DETAILED DESCRIPTION:
UCPVax study is a prospective multicenter phase I/II study: 54 patients with metastatic NSCLC will be enrolled in 5 centers in France.

A translational research program will be performed to better define the eligibility criteria and predictive biomarkers needed for randomized phase II and Phase III trials.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Histologically or cytologically confirmed NSCLC (adenocarcinoma, squamous cell carcinoma, large cell carcinoma, undifferentiated carcinoma or other)
* Stage IIIB not amenable to radiotherapy or stage IV cancer according to the TNM classification (7th edition) or recurrent NSCLC after surgery not amenable to loco-regional therapy.
* Pre-treated with at least 2 or 3 lines of treatment (including immunotherapy). Chemoradiation for stage IIIB disease is considered as one treatment line.
* At least one measurable lesion by CT scan or MRI based on RECIST criteria version 1.1
* Performance status 0 or 1 on the ECOG scale
* Life-expectancy > 3 months
* Adequate hematological, hepatic, and renal function

Exclusion Criteria:

* Prior history of other malignancy except for: basal cell carcinoma of the skin, cervical intra-epithelial neoplasia and other cancer curatively treated with no evidence of disease for at least 5 years
* Symptomatic brain metastases. Patients with controlled brain metastases after radiation therapy or with asymptomatic brain metastases may be included.
* History of active autoimmune diseases (lupus, rheumatoid arthritis, inflammatory bowel disease…)
* Patients under chronic treatment with systemic corticoids or other immunosuppressive drugs (prednisone or prednisolone ≤ 10 mg/day is allowed) - - Positive serology for Human Immunodeficiency Virus (HIV) or Hepatitis C virus (HCV); presence in the serum of the antigens HBs
* Participation in a clinical study with an investigational product within 4 weeks prior to the start of the study treatment
* Pregnancy or lactating patients.
* Patients with any medical or psychiatric condition or disease,
* Patients under guardianship, curatorship or under the protection of justice.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-04-20 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) of UCPVax (phase I) | until day 57 after the first vaccination
  The following adverse events graded according to CTCAE v 4.03 will be classified as DLTs :
  * Hematologic:
    * Grade 4 neutropenia (ANC <0.5 x 109/L) lasting >5 days;
    * Febrile neutropenia (defined as neutropenia ≥Grade 3 [ANC <1000 cells/mm3] and a body temperature ≥38.5°C);
    * Grade ≥3 thrombocytopenia (<50.0 - 25.0 x 109/L) with bleeding;
    * Grade 4 thrombocytopenia (<25.0 x 109/L) >5 days;
    * Grade 4 anemia (hemoglobin <6.5 g/dL or 4.0 nmol/L);
  * Non-hematologic:
    o Grade ≥3 toxicities, except for alopecia and those grade 3 events that respond to treatment (eg. grade 3 nausea, vomiting, diarrhea that responds to standard medical supportive care within 48 hours will not be considered a DLT).
  * Immune system disorder:
    * Grade ≥2 allergic reaction (except for local reaction at the injection site : grade ≥ 3)
    * Grade ≥2 autoimmune disease (colitis, thyroidis…)
    * Grade ≥2 cytokine release syndrome (nausea, headache, tachycardia, hypotension, rash and shortness of breath)
Dose-related immunogenicity (phase II) | at day 73
  Antigen-specific T cell responses measured using IFN-gamma ELISPOT.

SECONDARY OUTCOMES:
Tumor response | every 8 weeks up to 15 months
  Tumor response evaluated per RECIST v1.1.
Progression-free survival (PFS) | through study completion, an average of 2 years
  delay from the date of inclusion to the disease progression (RECIST) or death from any cause whichever occurs first,
Overall survival (OS) | through study completion, an average of 2 years
  delay from the date of inclusion to death from any cause.
Health related Quality of Life (QoL) | through study completion, an average of 2 years
  HrQoL will be assessed using EORTC QLQ-C30 and LC13 modules specific to lung cancer
Adverse Events according to NCI CTCAE v.4.03 | through study completion, an average of 2 years

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - Centre Hospitalier Régional Universitaire de Besançon, Besançon
  - Centre Georges François Leclerc, Dijon
  - Hôpital Emile Muller, Mulhouse
  - St Louis Hospital, Paris
  - Hôpitaux Universitaires de Strasbourg, Strasbourg

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galaine J, Borg C, Godet Y, Adotevi O. Interest of Tumor-Specific CD4 T Helper 1 Cells for Therapeutic Anticancer Vaccine. Vaccines (Basel). 2015 Jun 30;3(3):490-502. doi: 10.3390/vaccines3030490. PMID 26350591
- [Background] Dosset M, Godet Y, Vauchy C, Beziaud L, Lone YC, Sedlik C, Liard C, Levionnois E, Clerc B, Sandoval F, Daguindau E, Wain-Hobson S, Tartour E, Langlade-Demoyen P, Borg C, Adotevi O. Universal cancer peptide-based therapeutic vaccine breaks tolerance against telomerase and eradicates established tumor. Clin Cancer Res. 2012 Nov 15;18(22):6284-95. doi: 10.1158/1078-0432.CCR-12-0896. Epub 2012 Oct 2. PMID 23032748
- [Background] Godet Y, Fabre E, Dosset M, Lamuraglia M, Levionnois E, Ravel P, Benhamouda N, Cazes A, Le Pimpec-Barthes F, Gaugler B, Langlade-Demoyen P, Pivot X, Saas P, Maillere B, Tartour E, Borg C, Adotevi O. Analysis of spontaneous tumor-specific CD4 T-cell immunity in lung cancer using promiscuous HLA-DR telomerase-derived epitopes: potential synergistic effect with chemotherapy response. Clin Cancer Res. 2012 May 15;18(10):2943-53. doi: 10.1158/1078-0432.CCR-11-3185. Epub 2012 Mar 8. PMID 22407833
- [Background] Godet Y, Dosset M, Borg C, Adotevi O. Is preexisting antitumor CD4 T cell response indispensable for the chemotherapy induced immune regression of cancer? Oncoimmunology. 2012 Dec 1;1(9):1617-1619. doi: 10.4161/onci.21513. PMID 23264913
- [Background] Adotevi O, Dosset M, Galaine J, Beziaud L, Godet Y, Borg C. Targeting antitumor CD4 helper T cells with universal tumor-reactive helper peptides derived from telomerase for cancer vaccine. Hum Vaccin Immunother. 2013 May;9(5):1073-7. doi: 10.4161/hv.23587. Epub 2013 Jan 28. PMID 23357860
- [Result] Adotevi O, Vernerey D, Jacoulet P, Meurisse A, Laheurte C, Almotlak H, Jacquin M, Kaulek V, Boullerot L, Malfroy M, Orillard E, Eberst G, Lagrange A, Favier L, Gainet-Brun M, Doucet L, Teixeira L, Ghrieb Z, Clairet AL, Guillaume Y, Kroemer M, Hocquet D, Moltenis M, Limat S, Quoix E, Mascaux C, Debieuvre D, Fagnoni-Legat C, Borg C, Westeel V. Safety, Immunogenicity, and 1-Year Efficacy of Universal Cancer Peptide-Based Vaccine in Patients With Refractory Advanced Non-Small-Cell Lung Cancer: A Phase Ib/Phase IIa De-Escalation Study. J Clin Oncol. 2023 Jan 10;41(2):373-384. doi: 10.1200/JCO.22.00096. Epub 2022 Sep 7. PMID 36070539
- [Derived] Laheurte C, Boullerot L, Ndao B, Malfroy M, Queiroz L, Guillaume P, Loyon R, Seffar E, Gravelin E, Renaudin A, Jacquin M, Meurisse A, Vernerey D, Ghiringhelli F, Godet Y, Genolet R, Jandus C, Borg C, Adotevi O. UCPVax, a CD4 helper peptide vaccine, induces polyfunctional Th1 cells, antibody response, and epitope spreading to improve antitumor immunity. Cell Rep Med. 2025 Jul 15;6(7):102196. doi: 10.1016/j.xcrm.2025.102196. Epub 2025 Jun 20. PMID 40543509